CLINICAL TRIAL: NCT07183046
Title: Impact of an Implementation Intention Planning Guide on Fecal Immunochemical Tests (FIT) Completion Rates
Brief Title: Implementation Intention Planning Guide for FIT Colon Cancer Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audrey H. Calderwood, Director, Comprehensive Gastroenterology Center; Professor of Medicine, Geisel School of Medicine and the Dartmouth Institute; Staff physician, Gastroenterology and Hepatology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY02002735
Record Dates: First submitted 2025-07-29; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-07

CONDITIONS: Fecal Immunochemical Test; Colorectal Cancer Screening

STUDY DESIGN:
Intervention Model Description: Participants will be grouped into intervention and control groups based on alternating weeks/months when they obtain their FIT throughout the study. These timelines will be designated before the initiation of the study with appropriate frequency of alternation to reduce variability between non-study conditions between the weeks/months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (FIT Standard of Care) (No Intervention): The Control Arm will receive the fecal immunochemical test (FIT) standard of care. Participants in this arm will be evaluated by their ordering provider about their eligibility and appropriateness for FIT for colorectal cancer screening. If appropriate, these participants will receive the FIT, instructions, and any other documentations always provided to participants receiving FIT in clinical practice. Any follow-up materials or communications with their provider will also follow FIT standard of care. They will not receive any additional document/implementation intention guide with their FIT.
- Intervention Arm (FIT Standard of Care with Implementation Intention Guide) (Experimental): The Intervention Arm will receive the fecal immunochemical test (FIT) standard of care and the implementation intention guide one-page document. Participants in this arm will be evaluated by their ordering provider about their eligibility and appropriateness for FIT for colorectal cancer screening. If appropriate, these participants will receive the FIT, instructions, and any other documentations always provided to participants receiving FIT in clinical practice. They will also receive the implementation intention guide being evaluated in this study. Any follow-up materials or communications with their provider will also follow FIT standard of care.
  Interventions: Behavioral: Implementation Intention Guide

INTERVENTIONS:
Behavioral: Implementation Intention Guide — The intervention is the addition of implementation intention guide document provided with the FIT. This is a one-page piece of paper that was developed by the investigator team and finalized with input/feedback from patient partners. The implementation intention guide includes instructions about the importance of developing a plan to complete FIT. It also includes fillable fields for participants to enter their plan for when to complete, where to store, when to return, and where to return their FIT. Participants will also be able to follow a QR code on the implementation intention guide document to a link to complete an anonymous, electronic version of the guide and share feedback on the intervention.
  Arms: Intervention Arm (FIT Standard of Care with Implementation Intention Guide)

SUMMARY:
Fecal immunochemical tests (FIT) are a primary method of screening for colorectal cancer (CRC). Implementation intention planning involves encouraging completion or eliminating barriers for the participant to make a plan to complete a behavior or activity. This randomized control study seeks to answer whether the addition of an implementation intention guide impacts behaviors when completing FIT screening. The primary objective includes determining if the implementation intention guide increases completion rate of screening FIT. The secondary objectives is whether this intervention decreases the lab sample rejection rate and reduces the duration between sample collection and laboratory receipt/evaluation of screening FIT.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) has a high incidence, burden of disease, and significant associated mortality.(1,2) Programs to screen for CRC have leveraged stool testing with the fecal immunochemical test (FIT), a non-invasive at home test with no inherent risks, as the primary method in many countries.(3) Advantages of screening with FIT include considerations of safety, simplicity, and cost. However, while this and other options are available for colorectal cancer screening, patient screening rates have still not achieved recommended 70-80% targets.(4) In order to increase colorectal cancer screening rates, various behavioral interventions (including screening reminders, mailed screening outreach, choice architecture) have been implemented with success.(5,6)

Implementation intention planning involves encouraging or eliminating barriers for the participant to make a plan and complete FIT. Prior examples found that touchscreen implementation intention planning increased CRC screening completion by 12%.(7) For FOBT specifically, implementation intention planning instructions increased completion by 1.2-6.6%.(8) However, pre-written tips about FIT related to barriers did not increase FIT completion.(9)

This study seeks to understand the impact of a simple implementation intention planning guide (one-page piece of paper) on increasing rates of successful completion of FIT for colorectal cancer screening. The implementation intention planning guide is a one-page document that encourages the patient to make concrete plans about completing FIT. This study will evaluate if this low-cost intervention improves the rate of successful completion and reduces the duration between sample collection and lab result.

While some versions of implementation intention planning for CRC screening have been evaluated and shown positive impact in CRC screening completion, this study is hoping to build on these findings to evaluate a simplified implementation intention guide for patients specific to FIT. If this intervention is found to improve completion, these significant findings would support future FIT programs with a simple intervention to improve community screening rates. If these interventions do not improve completion, this research will inform the need to pursue investment in evaluating other interventions to improve FIT screening rates.

Aim 1: To determine if inclusion of implementation intention guide in FIT increases 90-day completion rate of screening FIT.

Hypothesis 1: The inclusion of implementation intention guide in FIT will increase the 90-day completion rate of screening FIT by 7%.

Aim 2: To determine if inclusion of implementation intention guide with FIT reduces the duration between sample collection and laboratory receipt/evaluation of screening FIT.

Hypothesis 2: The inclusion of implementation intention guide in FIT will reduce the duration between sample collection and laboratory receipt/evaluation by 20% in number of days and increase the number of samples received in the clinically appropriate time window of screening FIT (reducing the sample rejection rate) by 20%.

References:

1. Siegel RL, Wagle NS, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2023. CA: A Cancer Journal for Clinicians. 2023/05// 2023;73(3):233-254. doi:10.3322/caac.21772
2. Araghi M, Soerjomataram I, Jenkins M, et al. Global trends in colorectal cancer mortality: projections to the year 2035. https://doi.org/10.1002/ijc.32055. International Journal of Cancer. 2019/06/15 2019;144(12):2992-3000. doi:https://doi.org/10.1002/ijc.32055
3. Young GP, Rabeneck L, Winawer SJ. The Global Paradigm Shift in Screening for Colorectal Cancer. Gastroenterology. 2019/03/01/ 2019;156(4):843-851.e2. doi:https://doi.org/10.1053/j.gastro.2019.02.006
4. Green BB. Colorectal Cancer Control: Where Have We Been and Where Should We Go Next? JAMA Intern Med. 2018/12/01/ 2018;178(12):1658. doi:10.1001/jamainternmed.2018.4627
5. Mehta SJ, Palat S, McDonald C, et al. A Randomized Trial of Choice Architecture and Mailed Colorectal Cancer Screening Outreach in a Community Health Setting. Clinical Gastroenterology and Hepatology: The Official Clinical Practice Journal of the American Gastroenterological Association. 2024/04/30/ 2024:S1542-3565(24)00390-2. doi:10.1016/j.cgh.2024.04.003
6. Deeds S, Schuttner L, Wheat C, et al. Automated Reminders Enhance Mailed Fecal Immunochemical Test Completion Among Veterans: a Randomized Controlled Trial. J GEN INTERN MED. 2024/01// 2024;39(1):113-119. doi:10.1007/s11606-023-08409-8
7. Greiner KA, Daley CM, Epp A, et al. Implementation Intentions and Colorectal Screening. American Journal of Preventive Medicine. 2014/12// 2014;47(6):703-714. doi:10.1016/j.amepre.2014.08.005
8. Neter E, Stein N, Barnett-Griness O, Rennert G, Hagoel L. From the Bench to Public Health. American Journal of Preventive Medicine. 2014/03// 2014;46(3):273-280. doi:10.1016/j.amepre.2013.11.008
9. Lo SH, Good A, Sheeran P, et al. Preformulated implementation intentions to promote colorectal cancer screening: A cluster-randomized trial. Health Psychology. 2014 2014;33(9):998-1002. doi:10.1037/a0033507

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75
* Cared for by primary care at General Internal Medicine Clinic, Dartmouth-Hitchcock Medical Center (Lebanon, NH), Dartmouth Hitchcock Clinics Heater Road Primary Care (Lebanon, NH), Dartmouth Hitchcock Clinics Lyme Primary Care (Lyme, NH), or White River Junction Veterans Affairs Medical Center (White River Junction, VT) OR eligible for FIT through VA Mailed FIT Program

Exclusion Criteria:

* none

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
FIT completion rate | Through study completion, approximately 12-18 months
  Percentage of participants who have completed, returned, and have received completed lab results for FIT 90 days following participant reception of FIT.

SECONDARY OUTCOMES:
Duration between FIT collection date and receipt by the laboratory | Through study completion, approximately 12-18 months
  Number of days from the participant FIT collection date (as reported by the participant on the FIT collection bottle) to the date the lab received the participant's FIT.
Rate of lab sample rejection | Through study completion, approximately 12-18 months
  Percentage of FIT samples rejected from the lab to not be appropriate for further evaluation (e.g., incorrect sampling/storage, expired test)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Dartmouth Hitchcock Clinics, Heater Road Primary Care, Lebanon, New Hampshire
  - Dartmouth-Hitchcock Medical Center, General Internal Medicine Clinic, Lebanon, New Hampshire
  - Dartmouth Hitchcock Clinics, Lyme Primary Care Clinic, Lyme, New Hampshire
  - White River Junction Veterans Affairs Medical Center, Primary Care Clinic, White River Junction, Vermont
  - White River Junction Veterans Affairs Medical Center, VA Mailed FIT Program, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No